CLINICAL TRIAL: NCT03049605
Title: Effects of Electromagnetic Therapy Versus Laser Therapy on Peripheral Neuropathy in Diabetic Patients
Brief Title: Effects of Electromagnetic Therapy Versus Laser Therapy on Peripheral Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014171
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes
Keywords: Neuropathies laser and magnetic therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Magnetic Field Therapy; Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: By randomization of participants recruitment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Magnetic Therapy (Experimental): Twenty five patient were exposed to low intensity pulsed magnetic therapy with a frequency of 200 Hertz and intensity of 50 Gauss for 30 minutes / session for 2 times per week for 3 months .
  Interventions: Device: Magnetic therapy
- Laser Therapy (Experimental): Twenty five patients were treated with 24 sessions of laser therapy at a rate of two sessions / week for three months. Each patient will be exposed to Helium neon infrared laser (850 nano-meter continuous wave mode from a comfortable prone lying position.
  Interventions: Device: laser therapy
- Medical therapy (Experimental): Fifteen patients were received only medical treatment .
  Interventions: Drug: Only medical treatment

INTERVENTIONS:
Device: Magnetic therapy — low intensity pulsed magnetic therapy with a frequency of 200 Hertz and intensity of 50 Gauss . Magnetic device will be applied on each patient from a comfortable supine lying position. After the connection of appliance to electrical supply, the actions of PEMF will be directed and adjusted over lumbar spine, hip regions and calf muscles of both lower limbs.
  Arms: Magnetic Therapy
Device: laser therapy — laser therapy of Helium neon infrared laser (850 nano-meter) was used in continuous wave mode from a comfortable prone lying position on the whole plantar surface of the foot and the lumbo-sacral area by four points, and two points laterally to the spine.
  Arms: Laser Therapy
Drug: Only medical treatment — Fifteen patients with diabetic peripheral neuropathy were treated with antidiabtic drugs and lyrica 150 milligram daily
  Other Names: Lyrica 150 milligram
  Arms: Medical therapy

SUMMARY:
This study are to:

* Evaluate effect of magnetic therapy on peripheral neuropathy in diabetic patients.
* Evaluate effect of laser therapy on peripheral neuropathy in diabetic patients.
* Compare effects of magnetic therapy with that of laser therapy on peripheral neuropathy in diabetic patients.

DETAILED DESCRIPTION:
Sixty- five male and female diabetic patients with peripheral neuropathy will be selected to participate in this study. They will be equally divided into two groups Group-I: Twenty five patient with diabetic peripheral neuropathy will be exposed to low intensity pulsed magnetic therapy Group-II: Twenty five patients with diabetic peripheral neuropathy will be exposed for 24 treatment sessions of laser therapy Group-III 15 patient received only medical treatment

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients with peripheral neuropathy will be selected to participate in this study.
* Their age ranges from 35 to 65 years old.
* All patients under medical control (optimal blood glucose). such as analgesic medications (e.g. opiates, anti-depressants, anticonvulsants and diabetic drugs to control blood glucose).

Exclusion Criteria:

* Patients have DPN due to other causes than diabetes
* Ulcers in either foot
* Lack of blood sugar control
* Other nervous system impairments
* Visual problems
* Unstable medical conditions
* Pregnancy
* Metallic implants
* Alcohol or drug abuse.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01-25 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Motor and sensory conduction velocity of the lower limb nerves | 30-45 minutes
  it is used for measuring motor and sensory conduction velocity: For this purpose nerve conduction studies (NCSs) will be performed for all patients including evaluation of bilateral peroneal and tibia motor nerves and sural sensory nerves (Asad 2009). Patients with NCV from 33-48m /sec will be recruited in this study (Pericz and Cvetkovic 2006 , and Graak 2009). All measurement will be done at stander room temperature of 25 c. The skin temperature of the leg was maintained at 37ᴄ. (Asad et al 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Enas F. Alananey, PhD, Study Director — Associate professor university of Dammam

IPD SHARING:
Plan to Share IPD: No
The individuals date not shared but the final results comments will appear only

REFERENCES:
- [Result] Bosi E, Conti M, Vermigli C, Cazzetta G, Peretti E, Cordoni MC, Galimberti G, Scionti L. Effectiveness of frequency-modulated electromagnetic neural stimulation in the treatment of painful diabetic neuropathy. Diabetologia. 2005 May;48(5):817-23. doi: 10.1007/s00125-005-1734-2. Epub 2005 Apr 15. PMID 15834546
- See also: it is a scientific location — https://www.ncbi.nlm.nih.gov/pubmed?term=.+Effectiveness+of+frequency-modulated+electromagnetic+neural+stimulation+in+the+treatment+of+painful+diabetic+neuropathy.+Diabetologia.&TransSchema=title&cmd=detailssearch